CLINICAL TRIAL: NCT02364349
Title: A Comparative Study on Local Allergic Responses of Bee Venom and Essential Bee Venom Pharmacopuncture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: JS-CT-2015-01
Record Dates: First submitted 2015-01-28; First posted 2015-02-18 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Bee Venoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bee Venom (BV) group (Active Comparator): All subjects are injected with Bee Venom (BV, intervention), randomly assigned to the right or left forearm. Raw BV used dried BV prepared through collection from bee venom sacs and removal of impurities. The BV administration site on each subject was on the palmar side of the designated arm 5 cm below the middle of the elbow crease as it is convenient for observation and has high responsiveness. Pharmacopuncture sessions were also conducted in the morning for higher responsiveness.
  Interventions: Drug: Bee Venom (BV)
- essential Bee Venom (eBV) group (Experimental): All subjects are injected with essential Bee Venom (eBV, intervention), randomly assigned to the right or left forearm. eBV was prepared through the following methods: BV was collected from bee venom sacs and dried. LC/MS was used to analyze subdivisions of dried BV dissolved in purified water and passed through a sephadex G-25 column to collect histamine-free units. Collected units were filtered to eliminate allergenic substances including PLA2 of molecular weight 10 kDa or higher. The eBV administration site on each subject was on the palmar side of the designated arm 5 cm below the middle of the elbow crease as it is convenient for observation and has high responsiveness. Pharmacopuncture sessions were also conducted in the morning for higher responsiveness.
  Interventions: Drug: Essential Bee Venom (e-BV)

INTERVENTIONS:
Drug: Bee Venom (BV) — Raw Bee Venom
  Other Names: Bee Venom pharmacopuncture; Bee Venom injection
  Arms: Bee Venom (BV) group
Drug: Essential Bee Venom (e-BV) — Bee venom without Hyaluronidase, Lysophospholipase, α-D-glucosidase, PLA2, Adolapin
  Other Names: Essential Bee Venom pharmacopuncture; Essential Bee Venom injection
  Arms: essential Bee Venom (eBV) group

SUMMARY:
This double-blinded randomized clinical trial investigates any differences in allergic responses elicited by Bee Venom (BV) and Essential Bee Venom (eBV).

DETAILED DESCRIPTION:
This double-blinded randomized clinical trial investigates difference in allergic responses elicited by Bee Venom (BV) and Essential Bee Venom (eBV). Twenty healthy volunteers aged 20-40 years were randomly allocated to the 2 groups and administered eBV and BV on left and right forearm, respectively, in accordance with group allocation. Physician, participant, and outcome assessor were blinded to group allocation. Local pain, swelling, itching, redness, wheals and adverse reactions were recorded by timepoint before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with no prior exposure to bee venom treatment
* Healthy individuals of both genders, 20 to 39 years old
* Individuals able to communicate their thoughts
* Voluntary participants who have provided written consent

Exclusion Criteria:

* Individuals on medications for chronic diseases (i.e. hypertension, hyperlipidemia)
* Individuals with past history of allergic dermatitis
* Individuals with past history of adverse events following bee stings
* Individuals with symptoms of common cold
* Individuals with fear of bee venom intervention or those who refuse to participate

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) on Pain | 0.5 hours after intervention
  Visual Analog Scale on Pain
Wheal and erythema | 24 hours after intervention
  traced on adhesive, transparent films and measured with 0.01mm calipher
Visual Analog Scale(VAS) on Pain | 48 hours after intervention
  Visual Analog Scale on Pain

SECONDARY OUTCOMES:
Visual Analog Scale(VAS) on Pain | 0, 2, 6, 24, 72, 96, 120, 144 hours after intervention
  Visual Analog Scale on Pain,
Visual Analog Scale(VAS) for Wheal response | 0,0.5, 2, 6, 24, 48, 72, 96, 120, 144 hours after intervention
  Wheal response
Visual Analog Scale(VAS) for Skin irritation | 0,0.5, 2, 6, 24, 48, 72, 96, 120, 144 hours after intervention
  Skin irritation
Wheal and erythema | 0, 0.5, 6, 24, 72 hours after intervention
  traced on adhesive, transparent films and measured with 0.01mm calipher
Adverse events | 0, 6, 24, 72 hours after intervention
  General skin irritation, Heat flush, Nausea, Vomiting, Pain, Headache, Dizziness, Fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Shik SHIN, MD, Study Chair — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No